CLINICAL TRIAL: NCT06939439
Title: Circulating Tumor DNA Monitoring for Postoperative Adjuvant Therapy Decision-Making in Stage III Gastric Cancer: A Prospective, Multicenter, Randomized Controlled Phase III Clinical Trial
Brief Title: Using ctDNA to Guide Treatment Decisions for Stage III Gastric Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: First Affiliated Hospital of Suzhou Medical College (Other); The Affiliated Hospital of Xuzhou Medical University (Other); Nanjing Gaochun People's Hospital (Other); The Affiliated Jiangning Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hao Xu, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLAYMORE
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Gastric Cancer Stage III
MeSH Terms: conditions — Stomach Neoplasms | interventions — tislelizumab

STUDY DESIGN:
Intervention Model Description: This randomized, controlled phase III clinical trial employs a parallel assignment model, where participants are allocated to one of two distinct treatment groups based on their postoperative ctDNA-MRD status. Patients with ctDNA-MRD positivity will be randomly assigned in a 1:1 ratio to either the trial arm (receiving tislelizumab combined with standard SOX chemotherapy) or the control arm (receiving SOX chemotherapy alone). The trial arm will receive tislelizumab administered at 200 mg intravenously every 3 weeks for 1 year, alongside 6-8 cycles of SOX chemotherapy (oxaliplatin 130 mg/m² intravenously every 3 weeks, plus tegafur based on body surface area orally twice daily for 14 days every 3 weeks). The control arm will receive SOX chemotherapy alone for 6-8 cycles. Patients with ctDNA-MRD negativity will receive standard SOX chemotherapy without randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tislelizumab + SOX Chemotherapy (Experimental): Patients in this group will receive tislelizumab (200 mg IV every 3 weeks for 1 year) in combination with SOX chemotherapy (oxaliplatin 130 mg/m² IV every 3 weeks and tegafur based on body surface area orally twice daily for 14 days every 3 weeks).
  Interventions: Drug: Tislelizumab + SOX Chemotherapy
- SOX Chemotherapy Alone (Active Comparator): Patients in this group will receive standard SOX chemotherapy alone (oxaliplatin 130 mg/m² IV every 3 weeks and tegafur based on body surface area orally twice daily for 14 days every 3 weeks).
  Interventions: Drug: SOX Chemotherapy

INTERVENTIONS:
Drug: Tislelizumab + SOX Chemotherapy — The intervention in this study involves the use of tislelizumab, a humanized IgG4 anti-PD-1 monoclonal antibody, in combination with the standard SOX chemotherapy regimen for postoperative adjuvant therapy in patients with stage III gastric or gastroesophageal junction adenocarcinoma who are ctDNA-MRD positive. Tislelizumab is administered at a dose of 200 mg intravenously every 3 weeks for a total duration of 1 year, alongside 6-8 cycles of SOX chemotherapy. The SOX regimen includes oxaliplatin (130 mg/m² intravenously every 3 weeks) and tegafur, with the dose of tegafur determined based on body surface area and administered orally twice daily for 14 days every 3 weeks.
  Arms: Tislelizumab + SOX Chemotherapy
Drug: SOX Chemotherapy — The control group will receive standard SOX chemotherapy alone, serving as an active comparator to evaluate the incremental benefit of adding tislelizumab. This design ensures a rigorous comparison while maintaining alignment with current standard-of-care practices.
  Arms: SOX Chemotherapy Alone

SUMMARY:
The goal of this randomized, controlled phase III clinical trial is to evaluate whether combining Tislelizumab with standard SOX chemotherapy improves disease-free survival (DFS) compared to chemotherapy alone in patients with stage III gastric or gastroesophageal junction adenocarcinoma who are ctDNA-MRD positive after surgery. The study will enroll 416 patients across multiple centers and will compare outcomes between two groups: patients receiving tislelizumab plus SOX chemotherapy and those receiving standard SOX chemotherapy alone. The primary questions to be addressed are whether the combination therapy improves 1-year DFS rates and whether it demonstrates an acceptable safety profile. Participants will provide tissue and blood samples for ctDNA-MRD testing, undergo postoperative adjuvant therapy (chemotherapy ± immunotherapy), and complete regular follow-up visits to monitor treatment response and safety. The trial will assess key outcomes, including DFS, overall survival (OS), and ctDNA clearance rates, to determine the clinical benefit and safety of tislelizumab in this population.

ELIGIBILITY:
Inclusion Criteria:

Histological or Cytological Confirmation: Patients must have a confirmed diagnosis of stage III gastric or gastroesophageal junction adenocarcinoma (according to the 8th edition of the American Joint Committee on Cancer (AJCC) staging system) based on histological or cytological examination.

Surgical Resection: Patients must have undergone D2 or more extensive lymph node dissection surgery, with available tumor tissue samples. Patients who received neoadjuvant therapy prior to surgery are excluded.

Age: Patients must be between 18 and 75 years of age. General Condition: Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.

Informed Consent: Patients must be able to understand the study protocol and voluntarily participate in the study, providing written informed consent.

Compliance: Patients must demonstrate good compliance, willingness to adhere to the treatment regimen specified in the study protocol, and ability to provide blood samples at designated time points.

Clinical Data: Patients must have complete imaging and pathological clinical data available.

Life Expectancy: Patients must have an expected survival of more than 3 months. Organ and Marrow Function: Patients must have adequate organ and bone marrow function.

Exclusion Criteria:

Inability to Confirm Diagnosis: Patients who cannot be confirmed as having primary stage III gastric or gastroesophageal junction adenocarcinoma through histological or cytological examination.

Inability to Receive Treatment: Patients who are unable to receive immune checkpoint inhibitors or SOX chemotherapy.

Inability to Comply with Follow-up: Patients who are unable to adhere to the predetermined clinical follow-up schedule.

Inability to Accept Study Protocol: Patients who cannot accept the treatment regimen specified in the study protocol.

Inability to Provide Efficacy Assessment: Patients who cannot undergo or provide designated efficacy assessment methods such as CT scans.

Autoimmune Diseases: Patients with a history of autoimmune diseases. Psychiatric or Substance Abuse Issues: Patients with a history of substance abuse that cannot be discontinued or those with psychiatric disorders, or any severe and/or uncontrolled medical conditions.

Severe Comorbidities: Patients with any severe comorbidities that, in the investigator's judgment, may jeopardize patient safety or completion of the study.

Pregnancy or Breastfeeding: Pregnant or breastfeeding women. Prior Neoadjuvant Therapy: Patients who received neoadjuvant therapy prior to surgery or intraoperative chemotherapy infusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
disease-free survival (DFS) | 1 year

SECONDARY OUTCOMES:
overall survival(OS) | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital with Nanjing Medical Unviersity, Nanjing, Jiangsu, China